CLINICAL TRIAL: NCT01533142
Title: Bariatric Surgery on the West Coast of Norway (Vestlandet): Prospective Study of Overweight People Undergoing Bariatric Surgery
Brief Title: Bariatric Surgery on the West Coast of Norway (Vestlandet)
Acronym: FatWest
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Helse Fonna (Other)
Collaborators: Helse Forde (Other); Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Bjørn Gunnar Nedrebø, MD, PhD, MD, PhD, Helse Fonna
Other Study IDs: 2010/3287
Record Dates: First submitted 2012-02-09; First posted 2012-02-15 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Weight Loss; Diabetes Mellitus; Urinary Incontinence
Keywords: lipids
MeSH Terms: conditions — Weight Loss; Diabetes Mellitus; Urinary Incontinence | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine and biopsi from fat
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- surgical methods: Different methods are used among hospitals in Helse-Vest, and this allows us to compare different clinical and biological effects following bariatric surgery different methods) among a homogeneous population in the western part of Norway (Vestlandet
  Interventions: Procedure: Bariatric surgery
- Morbid obesity
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Patients will be treated with one of two bariatric procedure::
  sleeve gastrectomy or gastric bypass
Procedure: Bariatric surgery — Surgical methods vary between hospitals: Voss: sleeve gastrectomy, Haugesund: gastric bypass (Roux-en Y),SUS: gastric bypass (Roux-en Y); Førde: biliopancreatic diversion with duodenal switch (BPD / DS) and sleeve gastrectomy

SUMMARY:
Bariatric surgery of morbid obesity was first located at Førde Central Hospital, but it is now an established treatment at several other hospitals in the health region (Voss Hospital (Helse Bergen), Haugesund Hospital (Helse Fonna) Stavanger University Hospital ((SUS) Helse Stavanger). Surgical methods vary between hospitals: Voss: sleeve gastrectomy, Haugesund: gastric bypass (Roux-en Y),SUS: gastric bypass (Roux-en Y); Førde: biliopancreatic diversion with duodenal switch (BPD / DS) and sleeve gastrectomy . The investigators have then in Helse-Vest a unique opportunity to examine the various clinical and metabolic effects from different surgical methods.

This project is part of the regional strategic research initiative in the Helse Vest

DETAILED DESCRIPTION:
Primary endpoints for the study are weight loss and self-reported quality of life (QoL) evaluated by Short Form (SF)-36 and Impact of Weight Wed Quality of Life-Lite (IWQOL-Lite)) Our hypothesis is that patients operated with RYGBP (Roux A-Y Gastric Bypass) and BPD / DS (biliopancreatic diversion with duodenal switch) have the same weight and same QoL after 5 years of follow-up as patients treated with gastric sleeve (laparoscopic gastric sleeve (LSG)) We will also compare the groups with respect to a number of secondary endpoints

400 patients (approximately 100 patients / institution) will be included in the main study. Some of the programs that run on secondary endpoints will be conducted separately under study at each hospital. These studies will be reported in separate articles.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes 18-60 years old
* Patients with morbid obesity that is applied to the bariatric surgery.
* Signed informed consent

Exclusion Criteria:

* Patients who become pregnant in the follow-up period will not continue in the study but the data will be treated as lost too follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Both sexes 18-60 years old Patients with morbid obesity that is applied to the bariatric surgery. Signed informed consent
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
weight loss | From 1 year and up to 5 years

SECONDARY OUTCOMES:
remission of diabetes mellitus type 2 | from 1 year up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Helse-Fonna, Haugesund, Haugesund, Norway

REFERENCES:
- [Derived] Grymyr LMD, Nadirpour S, Gerdts E, Nedrebo BG, Matre K, Cramariuc D. Long-Term Trajectories of Left Heart Geometry, Mechanics, and Oxygen Demand After Bariatric Surgery. Circ Heart Fail. 2025 May;18(5):e012367. doi: 10.1161/CIRCHEARTFAILURE.124.012367. Epub 2025 Apr 7. PMID 40190274
- [Derived] Grymyr LMD, Mellgren G, McCann A, Gerdts E, Meyer K, Nadirpour S, Ferno J, Nedrebo BG, Cramariuc D. Preoperative risk factors associated with left ventricular dysfunction after bariatric surgery. Sci Rep. 2024 Jan 25;14(1):2173. doi: 10.1038/s41598-024-52623-1. PMID 38273044
- [Derived] Grymyr LMD, Nadirpour S, Gerdts E, Nedrebo BG, Hjertaas JJ, Matre K, Cramariuc D. One-year impact of bariatric surgery on left ventricular mechanics: results from the prospective FatWest study. Eur Heart J Open. 2021 Aug 20;1(2):oeab024. doi: 10.1093/ehjopen/oeab024. eCollection 2021 Sep. PMID 35919265
- [Derived] Grymyr LMD, Nadirpour S, Gerdts E, Nedrebo BG, Hjertaas JJ, Matre K, Cramariuc D. Left ventricular myocardial oxygen demand and subclinical dysfunction in patients with severe obesity referred for bariatric surgery. Nutr Metab Cardiovasc Dis. 2021 Feb 8;31(2):666-674. doi: 10.1016/j.numecd.2020.10.009. Epub 2020 Oct 17. PMID 33257189